CLINICAL TRIAL: NCT06622473
Title: Experimental Evaluation of the Virtual Eggs Test on Stroke Participants
Acronym: VET_STROKE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Unknown)
Responsible Party: Principal Investigator, Francesca Cecchi, MD, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VirtualEggTest_STROKE
Record Dates: First submitted 2024-09-26; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stroke group (Experimental): each participant will perform the VET, NHPT, Abilhand-ULA, and Motricity Index with their most affected hand, followed by the VET and NHPT with the less affected hand.
  Interventions: Device: hand dexterity assessement

INTERVENTIONS:
Device: hand dexterity assessement — Each participant will perform the VET, with their most affected hand, followed by the VET with the less affected hand.

SUMMARY:
The study protocol focuses on evaluating the Virtual Eggs Test (VET) as a tool for assessing hand dexterity and grip strength control in post-stroke patients. The study aims to validate the reliability and concurrent validity of the VET, comparing its outcomes with established tests like the Nine Hole Peg Test (NHPT), the Motricity Index, the Semmes-Weinstein Monofilament Test (SWMT), and the Abilhand-ULA questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants of both sexes and any ethnicity, aged 18 to 85 years.
* Post-stroke patients:

  * Participants who have experienced a first ischemic or hemorrhagic stroke.
  * Participants must be in the sub-acute phase (between 2 weeks and 6 months after the stroke) or the chronic phase (more than 6 months after the stroke).
  * Sufficient motor capabilities to perform motor tasks.
* Cognitive and language capabilities: Participants must have sufficient cognitive and language abilities to understand the experiment and follow instructions.
* Informed consent: Participants must provide signed informed consent after being fully informed about the study.

Exclusion Criteria:

* Visual or oculomotor impairments: Participants with significant visual or eye movement disorders.
* Comorbidities/disabilities:

  * Participants with conditions such as multiple sclerosis, Parkinson's disease, muscle tone disorders, or malignant neoplasms, which may interfere with the ability to understand or perform the protocol.
  * Cardiopulmonary or circulatory pathologies.
* Pregnancy or breastfeeding.
* Psychiatric comorbidities.
* Language barriers: Participants unable to adequately understand the Italian language.
* Lack of collaboration: Participants who cannot cooperate sufficiently with the study requirements.
* Substance use: Consumption of alcohol or diuretics before the tests.
* Motor function criteria:

  * Participants with a Motricity Index score of <19 for the pinch grip item.
  * A total upper limb Motricity Index score of <57.
  * Participants with a fixed contracture of the affected limb (Modified Ashworth Scale = 4).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Threshold from the Virtual Eggs Test (VET) | First Session (Test)
  This refers to the grip strength threshold required to avoid breaking fragile objects during the test. The VET measures the participant's ability to regulate grip strength and dexterity, with the threshold ranging from 1 to 20. Lower numbers indicate that less force is needed to break the object, reflecting greater control over fine motor skills.
Semmes-Weinstein Monofilament Test (SWMT) | First Session (Test)
  A test that measures tactile sensitivity by applying calibrated filaments to the skin. The pressure exerted by the filaments ranges from 0.07 to 300 grams, with lower values indicating greater sensitivity and higher values indicating reduced sensation. The range helps to detect sensory deficits in the hands post-stroke.
Motricity Index (MI) | First Sessione (Test)
  A clinical assessment used to evaluate strength in the upper limb. It involves scoring the patient's ability to perform specific movements on a scale from 0 to 100, where 0 indicates no movement and 100 represents normal strength. Scores between 57 to 100 suggest varying degrees of strength in the upper limb.
Nine Hole Peg Test (NHPT) | First Session (Test)
  A timed test that assesses manual dexterity. The participant is asked to place and remove nine pegs from holes as quickly as possible. The total time is recorded, typically ranging from 20 to 60 seconds depending on the severity of impairment. Lower times indicate better dexterity.
Abilhand-ULA | First Session (Test)
  A self-assessment questionnaire used to measure manual ability in daily activities for individuals with upper limb impairments. Scores range from 0 to 2 for each item, where 0 means the task is impossible, 1 means it is difficult, and 2 means the task can be performed easily.
Threshold from the Virtual Eggs Test (VET) | Second Session (Re-Test)
  This refers to the grip strength threshold required to avoid breaking fragile objects during the test. The VET measures the participant's ability to regulate grip strength and dexterity, with the threshold ranging from 1 to 20. Lower numbers indicate that less force is needed to break the object, reflecting greater control over fine motor skills.

SECONDARY OUTCOMES:
Feasibility of the VET in a clinical setting | First Session (Test)
  Measurement of the average test duration in minutes
Feasibility of the VET in a clinical setting | Second Session (Re-Test)
  Measurement of the average test duration in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Carlo Gnocchi ONLUS, Florence, Florence, Italy

IPD SHARING:
Plan to Share IPD: No